CLINICAL TRIAL: NCT01564693
Title: Neuroimaging of Hypothalamic Activity During Cancer Anorexia
Brief Title: Cancer Anorexia and the Central Nervous System
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Alessandro Laviano, MD, Associate Professor, University of Roma La Sapienza
Other Study IDs: FRFLAV
Record Dates: First submitted 2012-03-14; First posted 2012-03-28 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-07

CONDITIONS: Cancer Cachexia
Keywords: anorexia; cancer; hypothalamus; inflammation
MeSH Terms: conditions — Anorexia; Neoplasms; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- ANOREXIC CANCER PATIENTS: Nine lung cancer patients were diagnosed as anorexic based on the results obtained by the appetite assessment tools we used. These patients were studied by fMRI regarding the hypothalamic activity.
- NON-ANOREXIC CANCER PATIENTS: Four lung cancer patients were diagnosed as non-anorexic based on the results obtained by the appetite assessment tools we used. These patients were studied by fMRI regarding the hypothalamic activity.
- CONTROL GROUP: Two healthy volunteers with normal appetite were studied by fMRI regarding the hypothalamic activity.

SUMMARY:
The pathogenesis of cancer anorexia is complex and multifactorial. However, a number of consistent and robust evidence point to a prominent role for the central nervous system. In particular, the hyperactivation of the immune system, due to tumour growth, causes a systemic inflammatory response primarily mediated by pro-inflammatory cytokines. At the central level, inflammatory response profoundly alters the activity of the hypothalamic nuclei, which are involved in the regulation of energy homeostasis. In particular, pro-inflammatory cytokines inhibit prophagic neurons activity, while enhance the activation of the anorexigenic neurons. Although supported by compelling experimental evidence, it should be acknowledged that this pathogenic hypothesis has not been confirmed yet by human studies.

Aim of the present study is to determine the specific pattern(s) of the brain activation after assumption of a standard meal in both anorexic and non-anorexic cancer patients to reveal potential differences, which will be correlated with the levels of concurrently measured circulating pro-inflammatory cytokines. The results obtained would help in assessing the role of the central nervous system and, in particular of the hypothalamus, in the pathogenesis of cancer anorexia.

DETAILED DESCRIPTION:
After approval of the study protocol by the Ethical Committee of our Institution (Azienda Policlinico Umberto I, Sapienza University, Rome, Italy), 9 anorexic cancer patients, 4 non-anorexic cancer patients and 2 healthy individuals will be studied. The sample size is based on studies of neuroimaging already published and available on international journals.

Patients with confirmed cancer diagnosis will be enrolled before the initiation of any anti-cancer treatments. The presence/absence of anorexia will be investigated using a specific questionnaire (Cangiano et al., 1990) and a visual analogue scale (VAS). After an overnight fasting, blood samples will be collected from cancer patients and control subjects and interleukin(IL)-1, IL-6 and Tumor Necrosis Factor-α (TNF-α) levels will be measured by a commercially available ELISA kit.

On the same day, hypothalamic activation pattern(s) will be evaluated in patients and in control subjects by fMRI. After basal evaluation, all the groups will receive a standard oral meal, i.e., a 200 mL hypercaloric oral nutritional supplement providing 300 Kcal, and then a second fMRI scan will be performed. Using a computerized software, the average value of the grey for the hypothalamus will be calculated, and normalized for the one obtained in the basal condition, to obtain the percentage (%) of activation (or inhibition) of the hypothalamus.

Data obtained will be statistically analyzed using the t-Student and Bonferroni tests.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer patients at diagnosis

Exclusion Criteria:

* Patients treated with immunosuppressors, with concomitant wasting diseases (e.g. AIDS, trauma, end-stage renal disease)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients with confirmed cancer diagnosis before the initiation of any anti-cancer treatments will be enrolled. Nine anorexic cancer patients, 4 non-anorexic cancer patients and 2 healthy individuals will be studied.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-04; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Laviano, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Department of Clinical Medicine, Sapienza University of Rome, Rome, Italy, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- ANOREXIC CANCER PATIENTS: We evaluated 9 patients with lung cancer who met the inclusion criteria and were enrolled in the study. According to the protocol, the presence of anorexia was assessed by appetite assessment tools.
- NON-ANOREXIC CANCER PATIENTS: According to the protocol, we evaluated 4 patients with lung cancer who met the inclusion criteria and were enrolled in the study. According to the protocol, the absence of anorexia was assessed by appetite assessment tools.
- CONTROL GROUP: Two healthy volunteers were evaluated and included in the study as controls. Their appetite was normal, as assessed by appetite measurement tools.
Period: Overall Study
Arm/Group | ANOREXIC CANCER PATIENTS | NON-ANOREXIC CANCER PATIENTS | CONTROL GROUP
Started | 9 (Originally we planned to study 4 patients. We expanded to 9 to improve consistency of the results.) | 4 | 2 (Only 2 patients were found necessary to give statistical relevance to the patients' results.)
Completed | 9 | 4 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ANOREXIC CANCER PATIENTS: Based on the anorexia instruments that we used, we considered these patients as anorexic.
- NON-ANOREXIC CANCER PATIENTS: Based on the anorexia instruments that we used, we considered these patients as non-anorexic
- CONTROL GROUP: These were healthy subjects. 1 MD working at the Oncology Dept. , 1 family member of one of the patients enrolled.
- Total: Total of all reporting groups
Arm/Group | ANOREXIC CANCER PATIENTS | NON-ANOREXIC CANCER PATIENTS | CONTROL GROUP | Total
Number analyzed (Participants) | 9 | 4 | 2 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 1 | 3
  >=65 years | 7 | 4 | 1 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (9.4) | 76.25 (6.95) | 65 (7.1) | 71.66 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 7
  Male | 6 | 1 | 1 | 8
Region of Enrollment [Number; unit: participants]
  Italy | 9 | 4 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: ACTIVATION/NON ACTIVATION OF SPECIFIC BRAIN AREAS, EVALUATED BY FUNCTIONAL MAGNETIC RESONANCE
Description: We observed different BOLD signal in the region of the hypothalamus between the 3 groups. The BOLD signal and the activation/no activation areas were statistically analyzed by a specific statistical method (i.e., parametric mapping).
Time Frame: TIME 0 (BASELINE)
Measure: Mean (Standard Deviation); unit: BOLD
Groups:
- ANOREXIC CANCER PATIENTS: Patients revealed as anorexic were studied regarding BOLD signal activity by fMRI
- NON-ANOREXIC CANCER PATIENTS: Patients revealed as non-anorexic were studied regarding BOLD signal activity by fMRI
- CONTROL GROUP: Healthy subjects were studied regarding BOLD signal activity by fMRI
Arm/Group | ANOREXIC CANCER PATIENTS | NON-ANOREXIC CANCER PATIENTS | CONTROL GROUP
Number analyzed (Participants) | 9 | 4 | 2
BOLD | 585.57 (55.69) | 667.92 (33.18) | 511.22 (79.43)

ADVERSE EVENTS:
Groups:
- ANOREXIC CANCER PATIENTS: Nine patients were studied by fMRI before and after administration of a standard meal. The presence of serious adverse events (i.e., allergy, claustrophobia) were investigated. The presence of nausea and vomiting after the intake of the standard meal was also investigated.
- NON-ANOREXIC CANCER PATIENTS: Four patients were studied by fMRI before and after administration of a standard meal. The presence of serious adverse events (i.e., allergy, claustrophobia) were investigated. The presence of nausea and vomiting after the intake of the standard meal was also investigated.
- CONTROL GROUP: Two volunteers were studied by fMRI before and after administration of a standard meal. The presence of serious adverse events (i.e., allergy, claustrophobia) were investigated. The presence of nausea and vomiting after the intake of the standard meal was also investigated.
Arm/Group | ANOREXIC CANCER PATIENTS | NON-ANOREXIC CANCER PATIENTS | CONTROL GROUP
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/9 | 0/4 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes